CLINICAL TRIAL: NCT06989372
Title: Serratus Posterior Superior Intercostal Plane Block, Versus Erector Spinae Facial Plane Blocks A Comparative Study for Postoperative Pain Control and Opioid Consumption for Patient Undergoing Modified Radical Mastectomy Surgery
Brief Title: Serratus Posterior Superior Intercostal Plane Block, Versus Erector Spinae Facial Plane Blocks
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammed Shabayek, Lecturer of Anesthesia, ICU and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FMASU R68/2025
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-03

CONDITIONS: Breast Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (SP) (Active Comparator): serratus posterior superior block
  Interventions: Procedure: serratus posterior superior block
- Group II (ES) (Active Comparator): erector spinae block
  Interventions: Procedure: erector spinae block

INTERVENTIONS:
Procedure: serratus posterior superior block — patients were placed in the lateral decubitus position for SPSIPB. The blocks were performed under the guidance of ultrasonography (USG), a high-frequency linear probe (SonoSite HFL50x, 15-6 MHz, 55-mm broadband linear array, USA) transducer was placed at the level of the spine scapula in the transverse plane, and the upper medial border of the scapula, trapezius muscle, serratus posterior superior muscle (SPSM), 2nd and 3rd ribs were visualized. The ultrasound probe is rotated 90 degrees in a parasagittal orientation to identify the first rib. After its identification, the second and third ribs are confirmed. An 80 mm sono visible needle (type) was inserted in the caudocranial direction just medial to the scapula with the in-plane technique and driven between the 2nd and 3rd ribs targeting the inferior part of the SPSM. The target was confirmed by injecting the test dose with saline. Thirty ml of 0.25% bupivacaine was subsequently injected
  Arms: Group I (SP)
Procedure: erector spinae block — US-guided ESPB, a commonly performed interfascial plane block, was first defined by Forero et al. (21). In this technique, LA is injected in the plane between the erector spinae muscles and the thoracic transverse processes. Thus, multiple thoracic levels are anesthetized by the LA spreading in a craniocaudal direction. The transducer was then placed approximately 3 cm lateral to the midline parasagittally. The T5 transverse process and the erector spinae, rhomboid major, trapezius muscles were viewed (i.e., from deep to superficial). The block needle was advanced in a craniocaudal direction using an in-plane approach through the trapezius, rhomboid major, and erector spinae muscles. After establishing contact with the hyperechoic transverse process, 30 mL of 0.25% bupivacaine was injected in small aliquots after hydrodissection (2-3 mL, 0.9% NaCl) and checking for negative blood aspiration after every 5 mL of injection.
  Arms: Group II (ES)

SUMMARY:
Mastectomy is currently the most effective treatment for breast cancers in women. postoperative pain management carries a high degree of difficulty, as the breast has complex innervation involving the intercostal (T1-T7), superficial cervical plexus (supraclavicular nerves) and brachial plexus .While severe acute pain is observed in approximately 40% of post-mastectomy patients, moderate-to-severe pain is observed in almost one-third of them .

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* ASA classification I and II

Exclusion Criteria:

* age below 18 or above 65 years
* ASA classification III or more

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours post operatively
  The primary outcome is the total morphine consumption of the patient in the first 24 h postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No